CLINICAL TRIAL: NCT04262232
Title: Adaptation of Ca-HELP Intervention in Rural Geriatric Cancer Patient Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Maury Regional Medical Center (Other); Brown University (Other); National Institute on Aging (NIA) (NIH); Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-04020220; P30AG022845-16 (NIH)
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Results first posted 2023-03-13 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This is a single arm study in which all participants will be exposed to the intervention (Ca-HELP).
Masking Description: No masking due to this being a single arm study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ca-HELP (Experimental): This intervention arm will consist of six components: (1) Assessment of current knowledge, attitudes, and preferences; (2) clarification and correction of misconceptions about cancer pain control; (3) teaching of relevant concepts (education about cancer pain control); (4) planning (identifying goals of care, creating achievable goals of care, and creating strategies to communicate goals of care to providers and family members); (5) rehearsal of communication strategies using role play exercises; and (6) portrayal of learned skills (patient applies skills in visit with healthcare provider).
  Interventions: Behavioral: Adapted Ca-HELP for Geriatric Cancer Patients

INTERVENTIONS:
Behavioral: Adapted Ca-HELP for Geriatric Cancer Patients — Intervention group: This intervention will be informed by social-cognitive theory10-13 and modeled after the tailored education and coaching intervention (TEC) used for Ca-HELP previously and consists of six components: (1) Assessment of current knowledge, attitudes, and preferences; (2) clarification and correction of misconceptions about cancer pain control; (3) teaching of relevant concepts (education about cancer pain control); (4) planning (identifying goals of care, creating achievable goals of care, and creating strategies to communicate goals of care to providers and family members); (5) rehearsal of communication strategies using role play exercises; and (6) portrayal of learned skills (patient applies skills in visit with healthcare provider).

SUMMARY:
The Cancer Health Empowerment for Living without Pain (Ca-HELP) is an evidence-based communication tool that empowers and engages patients to communicate effectively with their physicians about pain. The Ca-HELP intervention is rooted in social-cognitive theory which posits that behavior change and maintenance depends largely on individuals' ability and self-efficacy to execute a specific behavior. Ca-HELP coaches patients to ask questions, make requests, and signal distress to their physicians in order to achieve improved pain control. Previous research indicates significant improvement among cancer patients in their self-efficacy to communicate about their pain to their oncologists and reductions in pain misconceptions and pain-related impairment. Although a promising tool among geriatric cancer patients, Ca-HELP is not currently designed for optimal dissemination in rural settings.

DETAILED DESCRIPTION:
Overall study objective:

The objectives of this Stage I pilot study are to 1) adapt Ca-HELP for use in rural settings, and 2) inform research and trial design choices by engaging community partners. Following the completion of formative tasks about this adaptive design approach, investigators will conduct an open trial to test the feasibility and acceptability of methods and procedures for later use on a large scale R01-level RCT.

Specific Aims:

Aim 1: To adapt the Ca-HELP intervention for use with older adults with cancer in rural settings. This intervention adaptation will be informed by: (1) social-cognitive theory;12,13 (2) mixed methods analysis; and (3) semi-structured interviews from key stakeholder groups including patients, caregivers, and providers and hospital administration staff in rural clinic settings.

Aim 2: To evaluate the feasibility and acceptability of the adapted Ca-HELP intervention among older adults with cancer in rural clinic settings.

Hypothesis 2a: To evaluate feasibility, ≥70% of participants will meet the benchmark for feasibility defined by participant retention and adherence to the intervention.

Hypothesis 2b: To evaluate acceptability, ≥70% of participants will meet the benchmark for acceptability defined by responses on self-report measures of perceived helpfulness, satisfaction, and impact.

Aim 3: To test the preliminary efficacy of the Ca-HELP intervention adaptation on older adults with cancer to improve pain self-management (primary outcome) as well as pain misconceptions; self-efficacy to communicate with their physicians regarding pain severity, pain-related impairment, and pain severity (secondary outcomes).

Hypothesis 3: We hypothesize that the intervention will reduce patients' pain misconceptions, pain-related impairment, and pain severity and improve pain self-management and self-efficacy to communicate about pain with their physicians.

For Aim 1, investigators will collect feedback from older adults with cancer (n=10 patients), their caregivers (n=10), and providers and staff working in rural clinic settings (n=10) to determine the appropriateness of this intervention framework and best methods for implementation (e.g., in person health coach, telephone-based, etc.). Following these formative tasks, Aims 2 and 3 will be achieved through an open trial in rural Tennessee to test the intervention with n=30 older (65 years+) cancer patients in rural clinics and assess outcomes at baseline, post-intervention, and three months post-intervention.

ELIGIBILITY:
Patient Inclusion Criteria:

* 65 years of age or older
* Diagnosed with cancer
* English speaking
* Reside in non-institutional, rural settings
* Receive care at community-based clinic in rural area
* Ability to provide informed consent
* Have identified an informal caregiver.

Patient Exclusion Criteria:

* Severe cognitively impairment (Short Portable Mental Status Questionnaire scores of <6);
* Receiving hospice at time of enrollment.

Caregiver eligibility criteria include the following

* The person (family member or friend) whom the patient indicates provides most of their informal care
* Able to provide informed consent.

Provider eligibility criteria:

-Currently works with geriatric cancer patients OR in a healthcare system serving this patient population. Providers will include social workers, nurses, oncologists, and healthcare administrators.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cary Reid, MD, PhD, Principal Investigator — Weill Medical College of Cornell University; Megan Shen, PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Maury Regional Medical Center, Columbia, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ca-HELP
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ca-HELP
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.0 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 24
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30
Insurance status [Count of Participants; unit: Participants]
  Insured | 30
  Not insured | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility (Aim 2), as Measured by Number of Subjects Accrued to the Study
Description: Number of subjects accrued
Time Frame: Two weeks post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Ca-HELP
Number analyzed (Participants) | 30
Participants | 30

2. Primary Outcome: Feasibility (Aim 2), as Measured by Number of Subjects to Complete the Intervention
Description: Number of subjects to complete intervention
Time Frame: Two weeks post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Ca-HELP
Number analyzed (Participants) | 30
Participants | 30

3. Primary Outcome: Acceptability (Aim 2), as Measured by Qualitative Feedback
Description: Semi-structured interview assessing perceived satisfaction, helpfulness, usability, and readability. This interview will be coded qualitatively for themes that assess these components for assessment of overall acceptability. Qualitative data was analyzed as number of subjects endorsing specific themes. Themes around usability and readability did not emerge from the semi-structured interviews, thus no data on usability or readability were available to analyze.
Time Frame: Two weeks post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Ca-HELP
Number analyzed (Participants) | 30
Participants
  Satisfaction (Liked participating in intervention) | 25
  Helpfulness (Stated intervention was helpful) | 30

4. Primary Outcome: Acceptability (Aim 2), as Measured by Helpfulness
Description: Likert scale item assessing perceived helpfulness. Likert scale from 1 (not at all helpful) to 5 (very helpful), with 5 indicating higher levels of acceptability.
Time Frame: Two weeks post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ca-HELP
Number analyzed (Participants) | 30
score on a scale | 4.8 (0.5)

5. Primary Outcome: Acceptability (Aim 2), as Measured by Satisfaction
Description: Likert scale item assessing perceived satisfaction. Likert scale from 1 (not at all satisfied) to 5 (very satisfied), with 5 indicating higher levels of acceptability.
Time Frame: Two weeks post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ca-HELP
Number analyzed (Participants) | 30
score on a scale | 4.7 (0.64)

6. Primary Outcome: Acceptability (Aim 2), as Measured by Usability
Description: Likert scale item assessing perceived usability by assessing how difficult the intervention content was to understand. Likert scale from 1 (not at all) to 5 (very much). The item was reverse scored so that 5 indicates higher levels of acceptability.
Time Frame: Two weeks post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ca-HELP
Number analyzed (Participants) | 30
score on a scale | 4.7 (1.02)

7. Primary Outcome: Acceptability (Aim 2), as Measured by Readability
Description: Yes/no items assessing perceived readability (wording was too complicated, ideas were too complicated, there was too much information, there was not enough information). Individual items will be summed to create a total readability score. Scores can range from 0 (no issues/ good readability) to 4 (poor readability). *Note these questions were only answered among participants who indicated that the intervention content was difficult to understand (eg, poor usability) by scoring >1 on the 1 to 5 Likert-scale of usability.
Time Frame: Two weeks post-intervention
Population: Only 3 out of 30 participants scored >1 on the Likert-scale item, indicating some difficulty understanding the intervention. Of those 3, no participants indicated yes or no to items assessing possible readability. As such, there was no data available to analyze for this outcome.
Arm/Group | Ca-HELP
Number analyzed (Participants) | 0

8. Primary Outcome: Change in Pain Self-management (Aim 3)
Description: Two items from the pain management subscale of the Chronic Pain Self-Efficacy scale. Items rated on a 5-point Likert scale (1 = not at all certain and 5 = extremely certain). Scores range from 2 (low self-management) to 10 (high self-management).
Time Frame: Baseline, two weeks post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ca-HELP
Number analyzed (Participants) | 30
score on a scale
  Baseline | 6.2 (1.97)
  Two weeks post-intervention | 8.0 (1.23)
Statistical Analysis 1: Comparison: Ca-HELP; Test type: Superiority; p = 0.0001, Paired t-test, two-sided; Mean Difference (Net) = -1.8, 95% CI 2-sided [-2.6 to -0.95] — Baseline value minus two weeks post-intervention value

9. Primary Outcome: Change in Pain Misconceptions (Aim 3)
Description: Assessed using the 11 items based on the short version of the Barriers Questionnaire. Items are rated on a five-point Likert scale (1=disagree very much, 5=agree very much). Scores range from 1 (low misconception) to 5 (high misconception) as an average across all 11 items.
Time Frame: Baseline, two weeks post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ca-HELP
Number analyzed (Participants) | 30
score on a scale
  Baseline | 2.9 (0.54)
  Two weeks post-intervention | 1.5 (0.32)
Statistical Analysis 1: Comparison: Ca-HELP; Test type: Superiority; p < 0.0001, Paired t-test, two-sided; Mean Difference (Net) = 1.4, 95% CI 2-sided [1.17 to 1.63] — Baseline value minus two weeks post-intervention value

10. Secondary Outcome: Treatment Fidelity as Measured by Number of Subjects for Which the Intervention Was Delivered With Fidelity
Description: Treatment fidelity will be assessed with a checklist that captures whether session content was delivered and appropriate techniques were utilized.
Time Frame: Two weeks post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Ca-HELP
Number analyzed (Participants) | 30
Participants
  Fidelity (8-item checklist on communication; eg, pacing, volume, intro to intervention) | 27
  Fidelity (10-item checklist on delivery of intervention content across all 5 modules) | 30

11. Secondary Outcome: Change in Self-efficacy for Communicating With Physicians About Pain Severity
Description: Assessed using the 5-item Perceived Efficacy in Patient-Physician Interactions scale as modified to refer to communication with oncologists. Items are rated on a five-point Likert scale (1=not at all confident, 5 = very confident). Scores range from 5 (low self-efficacy) to 25 (high self-efficacy).
Time Frame: Baseline, two weeks post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ca-HELP
Number analyzed (Participants) | 30
score on a scale
  Baseline | 20.3 (5.28)
  Two weeks post-intervention | 23.1 (2.85)
Statistical Analysis 1: Comparison: Ca-HELP; Test type: Superiority; p = 0.01, Paired t-test, two-sided; Mean Difference (Net) = -2.8, 95% CI 2-sided [-4.99 to -0.61] — Baseline value minus two weeks post-intervention value

12. Secondary Outcome: Change in Pain-related Impairment
Description: Measured using the 6-item Medical Outcomes Study (MOS) Pain Impairment Scale. Items are rated on a five-point likert scale (1=not at all, 5 = extremely). Scores can range from 6 (low pain impairment) to 30 (high pain impairment).
Time Frame: Baseline, two weeks post-intervention
Population: The data was not collected at two weeks post-intervention due to an error in assessment. Thus, data is not reported for the post-intervention time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ca-HELP
Number analyzed (Participants) | 30
score on a scale
  Baseline | 13.8 (6.58)
  Two weeks post-intervention: number analyzed (Participants) | 0

13. Secondary Outcome: Change in Pain Severity
Description: Assessed as the mean of the average and worst pain over the past two weeks on a 0 to 10 scale (0 = no pain and 10 = worst pain imaginable).
Time Frame: Baseline, two weeks post-intervention
Population: A total of 29 out of 30 participants data were analyzed because n=1 patient was missing post-intervention assessments for pain severity.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ca-HELP
Number analyzed (Participants) | 29
score on a scale
  Baseline | 3.7 (3.02)
  Two weeks post-intervention | 3.2 (2.76)
Statistical Analysis 1: Comparison: Ca-HELP; Test type: Superiority; p = 0.51, Paired t-test, two-sided; Mean Difference (Net) = 0.5, 95% CI 2-sided [-1.02 to 2.02] — Baseline value minus two weeks post-intervention value

ADVERSE EVENTS:
Time Frame: Adverse events were collected for up to 4 weeks (date of enrollment to date of post-intervention assessment completed).
Arm/Group | Ca-HELP
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-19): https://cdn.clinicaltrials.gov/large-docs/32/NCT04262232/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-19): https://cdn.clinicaltrials.gov/large-docs/32/NCT04262232/ICF_001.pdf